CLINICAL TRIAL: NCT06155968
Title: Evaluating The Quality of Recovery After Elective Cesarean Section Using ObsQoR-10, A Comparative Study Between Two Modalities for Pain Control.
Brief Title: Evaluating The Quality of Recovery After Elective Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Adham Haggag, Associate proffesor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: FMASU R310/2023
Record Dates: First submitted 2023-11-18; First posted 2023-12-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Quality of Recovery; Elective Cesarean Section; Quadratus Lumborum Block; Patient Controlled Analgesia
MeSH Terms: interventions — Passive Cutaneous Anaphylaxis

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCA group (Active Comparator): : the PCA pump will be connected in a separate cannula. The pump contains 0.5 mg nalbuphine/ ml. the basal rate is 5ml/h and lock out time is 10 min.
  Interventions: Drug: PCA
- QL block group (Active Comparator): . Patients will receive bilateral ultrasonography (USG) guided block with 20 ml of 0.25 % bupivacaine on each side. The block is performed by anaesthesia consultants having experience of 5 years in ultrasound guided blocks. The procedure will be performed using aseptic technique (gown, gloves, facemask and protective sheath for the ultrasound probe).
  The curvilinear probe (2 5 MHz, SonoSite Turbo M) is placed in the transverse axial plane just cranial to the iliac crest. The "shamrock sign" was visualised (viz., the transverse process (TP) of vertebra L4 is the stem, whereas the erector spinae muscle (ESM) posteriorly, quadratus lumborum (QL) muscle laterally and the psoas major (PM) muscle anteriorly represent the three leaves). The needle is introduced using an in plane technique from the posterior end of the transducer through the QL muscle. The target for injection is the fascial plane between the QL and PM muscles.
  Interventions: Procedure: QL block

INTERVENTIONS:
Procedure: QL block — The curvilinear probe (2 5 MHz, SonoSite Turbo M) is placed in the transverse axial plane just cranial to the iliac crest. The "shamrock sign" was visualised (viz., the transverse process (TP) of vertebra L4 is the stem, whereas the erector spinae muscle (ESM) posteriorly, quadratus lumborum (QL) muscle laterally and the psoas major (PM) muscle anteriorly represent the three leaves). The needle is introduced using an in plane technique from the posterior end of the transducer through the QL muscle. The target for injection is the fascial plane between the QL and PM muscles..
  Arms: QL block group
Drug: PCA — the PCA pump will be connected in a separate cannula. The pump contains 0.5 mg nalbuphine/ ml. the basal rate is 5ml/h and lock out time is 10 min
  Arms: PCA group

SUMMARY:
Adequately validated patient-reported outcome measures are available, which can assess recovery profiles following childbirth. This study will explore the effect of two different methods for pain management on the quality of recovery of pregnant women undergoing cesarean section

DETAILED DESCRIPTION:
* Type of Study: RCT
* Study Setting: Obstetric theatre at Ain Shams University Hospital
* Study Period :6 months

As per routine hospital practice, the pre-anesthetic assessment is performed, two 18 G peripheral cannula are inserted and 1 mg of granisetron and 50 mg of ranitidine are administered intravenously (IV) as premedications one hour before the operation, and 10 mL/kg of Ringer's lactate solution was infused for 15 minutes as a preload. All the study participants received a standard spinal anesthetic consisting of 10-12 mg of 0.5% hyperbaric bupivacaine.

The patients will be monitored using electrocardiography, non-invasive blood pressure measurement and pulse oximetry (SpO2). Spinal injection will be performed under aseptic technique in the sitting position at L3-L4 or L4-L5 intervertebral space using a 27-G Quincke needle.

The patients will be laid down in a supine position and oxygen therapy will be initiated at a rate of 6 L/min via a facemask throughout the procedure.

The level of sensory block will be confirmed using sensation to cold, the accepted level for initiation of the surgery will be at T4-5level.

The motor block will be monitored using Modified Bromage scale. The blood pressure, heart rate will be monitored. If the systolic blood pressure reduced to 20% below the baseline or less than 90 mmHg, 5 mg ephedrine was administered intravenously. Moreover, if the heart rate slowed to 50 beats/min or less, 0.5 mg atropine was administered intravenously.

After the completion of surgery, the sealed opaque envelope containing the group allocation was opened by the attending anaesthesia resident (who was not a part of the study) to decide the mode of analgesia the patient shall receive.

In group QL: The parturients will be positioned in left lateral decubitus position. The back is cleaned with chlorhexidine gluconate solution and is draped with sterile drapes. The block is given using 21 G, 100 mm long (B Braun Stimuplex®A) insulated blunt tip needles. Patients will receive bilateral ultrasonography (USG) guided block with 20 ml of 0.25 % bupivacaine on each side. The block is performed by anaesthesia consultants having experience of 5 years in ultrasound guided blocks. The procedure will be performed using aseptic technique (gown, gloves, facemask and protective sheath for the ultrasound probe).

The curvilinear probe (2 5 MHz, SonoSite Turbo M) is placed in the transverse axial plane just cranial to the iliac crest. The "shamrock sign" was visualised (viz., the transverse process (TP) of vertebra L4 is the stem, whereas the erector spinae muscle (ESM) posteriorly, quadratus lumborum (QL) muscle laterally and the psoas major (PM) muscle anteriorly represent the three leaves). The needle is introduced using an in plane technique from the posterior end of the transducer through the QL muscle. The target for injection is the fascial plane between the QL and PM muscles.

In the PCA group: the PCA pump will be connected in a separate cannula. The pump contains 0.5 mg nalbuphine/ ml. the basal rate is 5ml/h and lock out time is 10 min.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status classification ΙΙ; and scheduled for elective cesarean section using a low transverse Pfannenstiel incision with spinal anesthesia.

Exclusion Criteria:

* (1) major hepatic, renal, or cardiovascular disease; (2) local infection; (3) bleeding disorder; (4) any contraindication for spinal anesthesia; or (5) known allergy to any drug used in the study (6) refusal to participate in the study (7) BMI > 35 (8) had opioid dependence (9) chronic analgesic usage (10) inability to use patient controlled analgesia (PCA) device.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — parturient undergoing cesarean section
Enrollment: 128 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
ObsQor-10 score | 24 hours postoperative
  compare the total ObsQor-10 score in both groups to determine which pain management intervention yields a better outcome.

SECONDARY OUTCOMES:
validation of ObsQoR-10 | 24 hours
  psychometric validation of the ObsQoR-10 score in a subset of Egyptian women undergoing elective cesarean section.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university, Cairo, Egypt